CLINICAL TRIAL: NCT00006356
Title: A Randomized Phase III Study for the Treatment of Recurrent Epithelial Ovarian Cancer: Chemotherapy Alone Versus Chemotherapy Followed by Secondary Cytoreductive Surgery in Patients With a Treatment-Free Interval of More Than 12 Months
Brief Title: Chemotherapy With or Without Surgery in Treating Patients With Recurrent Ovarian Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-55963; EORTC-55963
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Cisplatin

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving a chemotherapy drug before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Randomized phase III trial to study the effectiveness of chemotherapy with or without surgery in treating patients who have recurrent epithelial ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare survival and progression free survival in patients with ovarian epithelial cancer after receiving treatment with chemotherapy with or without secondary cytoreductive surgery.
* Determine the toxicity of these treatment regimens in these patients.
* Determine the complications related to surgical treatment in these patients.
* Compare the quality of life in these patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to stage at initial diagnosis (early stage I-IIa vs advanced stage IIb-IV), length of interval from end of prior first line chemotherapy (1-2 years vs more than 2 years), response to first 3 courses of second line induction chemotherapy in this study (no change vs partial remission vs complete remission), number of measurable tumor lesions (1 vs more than 1), largest tumor size of recurrence (less than 5 cm vs 5 cm or more), and participating center.

Patients receive second line induction chemotherapy with either 3 courses of a 3-4 week regimen or 6 courses of a weekly regimen of platinum based (cisplatin or carboplatin) therapy. Patients with no change, partial remission, or complete remission are randomized to one of two treatment arms.

* Arm I: Patients undergo secondary cytoreductive surgery within 14 days of randomization. Within 8 weeks after the last preoperative chemotherapy course, patients continue platinum based chemotherapy every 3-4 weeks for at least 3 additional courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients continue platinum based chemotherapy for at least 3 additional courses as in arm I.

Quality of life is assessed at baseline; before the 4th or 6th course of chemotherapy or 1 week before surgery; after the 6th course of chemotherapy in the chemotherapy only arm OR before the 4th or 6th course of chemotherapy in the surgery arm; 2 months after chemotherapy or after the 6th course of chemotherapy in the surgery arm; and then every 6 months for up to 5 years.

Patients are followed every 3 months for 2 years, and then every 6 months for 3 years or until disease progression.

PROJECTED ACCRUAL: Approximately 700 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed recurrent ovarian epithelial cancer after first line chemotherapy, unless clear evidence of clinically progressive disease
* Must have received prior first line chemotherapy consisting of at least 4 courses of either cisplatin or carboplatin

  * At least 12 months since prior chemotherapy
* Measurable disease by clinical exam or diagnostic laparoscopy

  * At least one lesion greater than 1 cm in diameter
* No leptomeningeal or brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.25 times upper limit of normal (ULN)
* SGPT less than 2 times ULN

Renal:

* Creatinine less than 1.6 mg/dL OR
* Creatinine clearance greater than 40 mL/min

Other:

* No peripheral neurotoxicity greater than grade 2
* No psychological, familial, sociological, or geographical condition that would preclude study
* No complete bowel obstruction
* No other malignancy except adequately treated basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No more than 1 prior regimen of chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2000-08; Primary Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Favalli, MD, Study Chair — Ospedale Sta. Maria Delle Croci
Locations (1):
- Spedali Civili, Brescia, Italy